CLINICAL TRIAL: NCT03829696
Title: Alternative Provision of Medication Abortion Via Advance Provision
Brief Title: Advance Provision of Medication Abortion
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study is not proceeding at this time.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Daniel Grossman, Professor in Department of Obstetrics, Gynecology and Reproductive Sciences and Director of Advancing New Standards in Reproductive Health (ANSIRH), University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: A128753_02
Record Dates: First submitted 2019-01-09; First posted 2019-02-04 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Early Abortion
MeSH Terms: interventions — Mifepristone; Misoprostol; ulipristal acetate

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Non-pregnant women (Experimental): Participants will be provided Mifeprex® (oral mifepristone 200 mg) and misoprostol 800 mcg to be administered buccally (at 24-48 hours following mifepristone) or vaginally (as soon as 6 hours following mifepristone) if unintended pregnancy occurs during the study period and the participant would like to end of the pregnancy. Participants who test positive for pregnancy will consult with a study clinician over the phone prior to administering mifepristone and misoprostol, and will then attend an in-person follow-up visit.
  All participants will be provided with a single dose of ella® (ulipristal acetate emergency contraception 30 mg) by a clinician at the beginning of the study, as well as 6 AccuHome® midstream urine pregnancy tests.
  Interventions: Drug: Mifeprex® (Mifepristone 200 mg); Drug: Misoprostol 800 mcg; Drug: ella® (ulipristal acetate emergency contraception 30 mg); Diagnostic Test: AccuHome® Pregnancy OTC Test

INTERVENTIONS:
Drug: Mifeprex® (Mifepristone 200 mg) — Participants will receive Mifeprex® (mifepristone 800 mcg) from a clinician when they are not pregnant. Participants who have an unintended pregnancy during the study period and would like to have a medication abortion will consult with a clinician for an over-the-phone evaluation of contraindications and gestational age. Participants who take the medications will be evaluated again in-person at a subsequent follow-up visit.
Drug: Misoprostol 800 mcg — Participants will receive misoprostol from a clinician when they are not pregnant. Participants who have an unintended pregnancy during the study period would like to have a medication abortion will consult with a clinician for an over-the-phone evaluation of contraindications and gestational age. Participants who take the medications will be evaluated again in-person at a subsequent follow-up visit.
Drug: ella® (ulipristal acetate emergency contraception 30 mg) — Participants will receive one dose of ella (emergency contraception) from a clinician at the same time of receiving mifepristone and misoprostol, in case the participant should have unprotected intercourse or failed contraception and want to prevent unintended pregnancy.
Diagnostic Test: AccuHome® Pregnancy OTC Test — Participants will receive 6 AccuHome® pregnancy tests, which are midstream urine pregnancy tests and provide results within 3 minutes. Participants may request additional tests to be mailed to them by the study at any time.

SUMMARY:
This mixed-methods study follows a prospective cohort of participants receiving Mifeprex® (mifepristone) by a clinician in advance of a potential unintended pregnancy. Women participating in this study will be assessed by a clinician and provided Mifeprex® and misoprostol in a clinical setting. To assess acceptability of this service delivery model among participants, and feasibility of implementing a larger randomized controlled trial, the study will survey participants, evaluate any clinical outcomes recorded during clinical visits, and interview participants about their experiences participating in the study.

DETAILED DESCRIPTION:
The overarching goal of the project is to improve access to early abortion by reducing barriers that patients face obtaining services. Currently, patients are prescribed and receive Mifeprex® and misoprostol directly from a clinician, who evaluates patients for medical eligibility and contraindications. The Mifeprex® may be taken in the facility or at home, and the misoprostol is taken 24-48 hours later at home. The FDA recommends a follow-up visit, which can be over the phone.

The purpose of this study is to pilot test the model of advance provision of medication abortion (MAB). In this model, patients at risk of unintended pregnancy and with a desire to avoid pregnancy will be assessed by a clinician and provided counseling on pregnancy recognition and testing, as well as how to administer MAB at home. For this pilot study, only patients who have previously had a MAB will be included, since this population has reported the highest interest in the model, and they are also already familiar with how to use the medications. The clinician will provide Mifeprex® and misoprostol to the patient at the time of counseling in case the patient becomes pregnant and wants to terminate the pregnancy using the medications up to 10 weeks gestation. Patients will contact a study clinician for an over-the-phone assessment of eligibility for MAB, including assessment of gestational age, before self-administration of Mifeprex® and misoprostol, and then attend a follow-up visit with the clinician.

Patients will sign the Danco Patient Agreement Form prior to receiving the medication. Clinicians dispensing the medications will have signed the Prescriber Agreement Form, and the medications will be dispensed in a clinic or hospital. Study investigators will monitor participant activity through surveys throughout the study. Participants will be given clear instructions on study participation and returning unused medications in an appropriate time frame. Clinicians will also re-evaluate participants by telephone before they take the medications and evaluate them in person at a subsequent follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years old
* Speak and read English or Spanish
* Have female reproductive anatomy
* Report a history of regular menses (>24 and <38 days ) in the past 3 years (other than during pregnancy)
* Not currently pregnant and not desiring to be pregnant in the next year
* Report having had a medication abortion with mifepristone and misoprostol at some point in the past
* Hemoglobin ≥10 g/dL
* Do not report a history of ectopic pregnancy
* Do not report a history of a hemorrhagic disorder or currently taking anticoagulants (or plan to start taking anticoagulants during study period)
* Do not report a history of chronic adrenal failure
* Do not report a history of inherited porphyria
* Do not report an allergy to mifepristone or misoprostol
* Are not currently taking long-term corticosteroid therapy (>1 week)
* Considered at-risk for unintended pregnancy, defined as: those who report being sexually active (vaginal sex with a male); have not been told by a clinician that they cannot become pregnant; have not been sterilized and whose current sexual partner(s) has not been sterilized; who are not using a long-acting reversible contraceptive (LARC) or hormonal contraceptive; who use withdrawal, rhythm method, barrier method(s), spermicide, emergency contraception, and/or no method of contraception
* Say they would seek abortion if they became pregnant in the next year, and who do not express a preference for surgical abortion
* Willing and able to provide informed consent
* Have access to a working cellphone with them at the time of enrollment and are willing to receive calls and text messages from study staff
* Are planning to live within 25 miles of the study site for the 6 month study period

Exclusion Criteria:

* Younger than 18 years or older than 40 years
* Cannot speak and read English or Spanish
* Do not have female reproductive anatomy
* Report a history of irregular menses in the past 3 years
* Hemoglobin <10 g/dL
* Report a history of having an ectopic pregnancy
* Report a history of a hemorrhagic disorder or currently taking anticoagulants (or plan to start taking anticoagulants during study period)
* Report a history of chronic adrenal failure
* Report a history of inherited porphyria
* Report an allergy to mifepristone or misoprostol
* Currently taking long-term corticosteroid therapy (>1 week)
* Are not considered at-risk for unintended pregnancy, defined as: those who do not report being sexually active (vaginal sex with a male), have been told by a clinician they cannot become pregnant, have been sterilized or whose current sexual partner(s) has been sterilized, have an IUD or contraceptive implant in place, or currently taking hormonal contraception (oral contraceptive pills, patch or vaginal ring)
* Currently pregnant or desiring to become pregnant in the next year
* Have not had a medication abortion in the past
* Say if they became pregnant in the next year, they would not seek abortion or are unsure whether they would seek abortion; or who indicate a preference for surgical abortion Unwilling or unable to provide informed consent
* Do not have access to a working cellphone with them at the time of enrollment and are unwilling to receive calls or text messages from study staff
* Are not planning to live within 25 miles of the study site for the 6 month study period

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females at-risk of unintended pregnancy
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants satisfied with the advance provision model | Participants who do not take Mifeprex® will be surveyed 6 months following study enrollment. Participants who take Mifeprex® at any point during the 6 month study period will be surveyed one week after taking Mifeprex®.
  Proportion of participants who report being "somewhat satisfied" or "very satisfied" when asked "How satisfied are you with the advance provision model?"
Proportion of participants who are confident that they could use the abortion pills correctly if they got pregnant and decided to have an abortion using the advance provision model | Participants who do not take Mifeprex® will be surveyed 6 months following study enrollment. Participants who take Mifeprex® at any point during the 6 month study period will be surveyed one week after taking Mifeprex®.
  Proportion of participants who report "somewhat confident" or "completely confident" when asked "If you got pregnant and wanted an abortion in the next few months, how confident do you feel that you could use the abortion pills correctly?"
Proportion of participants who would recommend the advance provision model to a friend | Participants who do not take Mifeprex® will be surveyed 6 months following study enrollment. Participants who take Mifeprex® at any point during the 6 month study period will be surveyed one week after taking Mifeprex®.
  Proportion of participants who report "probably yes" or "definitely yes" when asked "Would you recommend getting the abortion pills in advance instead of going to a clinic to a friend?"

SECONDARY OUTCOMES:
Response rate to check-in and end-of-study surveys | End of the study, month 12
  The number of participants who respond to surveys will be monitored throughout the study period.
Number of participants who take Mifeprex® | End of study, month 12
  The number of participants who report taking Mifeprex® will be captured by clinical recording of study clinicians during over-the-phone assessments and follow-up visits, as well as data collected during check-in and end of study surveys.
Among participants who take Mifeprex®: Number of participants who take Mifeprex® and misoprostol correctly | End of study, month 12
  Correct use of medications will be assessed by the clinician at the time of follow-up care by a checklist of clinical criteria.
Among participants who take Mifeprex®: Gestational age at time of abortion | End of study, month 12
  Gestational age will be calculated by last menstrual period during the over-the-phone clinical evaluation with a study clinician. Ultrasound data will be analyzed if obtained.
Among participants who take Mifeprex®: Number of participants with an adverse event | Up to 6 weeks after reported use of Mifeprex®
  Number of participants who had a medical problem that required them to go to the hospital, emergency department or a doctor's office (other than regularly scheduled follow-up visit) after taking Mifeprex® and/or misoprostol.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Grossman, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] FDA (2016).
- [Background] Biggs MA, Ralph L, Raifman S, Foster DG, Grossman D. Support for and interest in alternative models of medication abortion provision among a national probability sample of U.S. women. Contraception. 2019 Feb;99(2):118-124. doi: 10.1016/j.contraception.2018.10.007. Epub 2018 Nov 15. PMID 30448203